CLINICAL TRIAL: NCT01308385
Title: Prediction and Characterization of Acute and Chronic Postoperative Pain - a Longitudinal Observational Study of the Relationship Between Experimental Pain Modulation and Clinical Postoperative Pain in Patients Undergoing Minimally Invasive Repair of Pectus Excavatum
Brief Title: Prediction and Characterization of Acute and Chronic Postoperative Pain
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MIRPEX-2
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Pain; Pain, Postoperative; Funnel Chest
MeSH Terms: conditions — Pain; Pain, Postoperative; Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with pectus excavatum
  Interventions: Other: Conditioned pain modulation

INTERVENTIONS:
Other: Conditioned pain modulation — When evaluating conditioned pain modulation, pressure pain threshold in the musculus quadriceps femoris act as test stimulus and 2 minutes cold pressor test (stirred ice and water) acts as the conditioning stimulus. The difference between pain thresholds before and after the cold pressor test is defined as the effect of CPM.

SUMMARY:
Despite enormous progress insufficient postoperative pain management remains a frequent problem in the early postoperative phase after surgery. Furthermore, the pain that persists after healing of the surgical wound is a large, but often unrecognized, clinical problem and it is estimated that 5-10% of those undergoing surgery will develop severe persistent pain leading to chronic disability and psychosocial distress.

Conditioned Pain Modulation (CPM), also known as the phenomenon "pain-inhibits-pain", is a reduction in pain somewhere on the body in response to the application of a second painful stimulus outside the painful area. In recent years, the CPM has been identified as a psycho-physical measure with clinical relevance in characterizing the individual's ability to modulate pain and consequently the individual's disposition to acquire painful conditions.

The purpose of this study is primarily to assess the relationship between CPM efficacy and clinical postoperative pain (postoperative pain intensity, use of analgesics, the intensity of secondary hyperalgesia and allodynia, and the incidence of persistent postoperative pain) associated with minimally invasive repair of pectus excavatum. In addition, the study aims at identifying other patient- and/or surgery-related factors affecting the course of postoperative pain.

Hypothesis:

- The greater the positive difference between the experimental pressure pain threshold (kPa) measured before and after application of a second painful stimulus (Cold Pressor Test), the lower the risk of developing persistent postoperative pain.

Secondary hypotheses

* The greater the positive difference between the experimental pressure pain threshold (kPa) measured before and after application of a different experimental painful stimulus (Cold Pressor Test) lower the pain intensity in the early postoperative period.
* The greater the positive difference between the experimental pressure pain threshold (kPa) measured before and after application of a different experimental painful stimulus (Cold Pressor Test), the shorter duration of early postoperative pain.
* The greater the positive difference between the experimental pressure pain threshold (kPa) measured before and after application of a different experimental painful stimulus (Cold Pressor Test), the lower the usage of epidural analgesia (mg / ml).
* The larger the positive difference between the experimental pressure pain threshold (kPa) measured before and after application of a different experimental painful stimulus (Cold Pressor Test) the lower consumption of oral analgesics (mg / day).
* Severe acute pain in the early postoperative period (postoperative days 0-3) is positively associated with the development of persistent postoperative pain (6 months postoperatively).
* Presence of preoperative pain and / or high postoperative use of analgesics and / or high pain intensity during the first 6-8 weeks postoperatively predicts pain 6 months postoperatively.
* The higher pain intensity and discomfort associated with brush-evoked allodynia and / or pinprick (Von Frey) secondary hyperalgesia the greater the risk for developing persistent postoperative pain (6 months postoperatively).
* High levels of preoperative catastrophizing (assessed on the day of admission) is related to the severity of acute pain (rated third postoperative day) and chronic pain (assessed 6 months postoperatively), even if controlled for depression and anxiety.
* The degree of preoperative positive and negative emotions (as assessed on the day of admission) is related to the degree of acute pain (rated third postoperative day) and chronic pain (assessed 6 months postoperatively) so that negative emotions are associated with high levels of pain, while positive feelings are related to low levels of pain.
* The study population does not differ significantly from the normal population in terms of personality traits (emotional reactions, extraversion, openness to experience, friendliness, conscientiousness).
* The study population does not experience a significant change in personality traits during the first 6 months after surgery.
* The quality of life and self-esteem is lower among patients who develop persistent postoperative pain compared with pain patients.
* Quality of life and self-esteem improve as a result of minimally invasive repair of pectus excavatum.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing minimally invasive repair of pectus excavatum
* Age > 15 years old

Exclusion Criteria:

* Previous thoracic surgery interventions
* Disorders affecting the central or peripheral nervous system
* Chronic pain (pain intensity assessed by numerical rating scale > 3)
* Inability to speak and understand Danish (instructions, questionnaires)
* Inability to understand and participate in experimental pain modulation
* Psychiatric disorders (ICD-10)
* A history of frostbite in the non-dominant upper limb
* Sores or cuts on non-dominant upper limb
* Cardiovascular disease
* A history of fainting and/or seizures
* Fracture in non-dominant upper limb
* Reynaud's phenomenon

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elective consequtive patients admitted for surgical correction of pectus excavatum
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Persistent postoperative pain | 6 months postoperatively
  Pain that develops and persists after minimally invasive repair of pectus excavatum. Other causes of pain (e.g. infection) and preoperatively defined painful conditions are are excluded.

SECONDARY OUTCOMES:
Pain intensity at rest | Daily for up to 42 days postoperatively, at 6 months follow-up
  Pain intensity is measured by means of an 11-point numerical rating scale with the verbal anchors "No pain" and "Worst pain imaginable"
Pain intensity when active | Daily for up to 42 days postoperatively, at 6 months follow-up
  Pain intensity is measured by means of an 11-point numerical rating scale with the verbal anchors "No pain" and "Worst pain imaginable"
Pain unpleasantness/discomfort at rest | Daily for up to 42 days postoperatively, at 6 months follow-up
  Pain unpleasantness/discomfort is measured by means of an 11-point numerical rating scale with the verbal anchors "No unpleasantness/discomfort" and "Worst unpleasantness/discomfort imaginable"
Pain unpleasantness/discomfort when active | Daily for up to 42 days postoperatively, at 6 months follow-up
  Pain unpleasantness/discomfort is measured by means of an 11-point numerical rating scale with the verbal anchors "No unpleasantness/discomfort" and "Worst unpleasantness/discomfort imaginable"
Pain location | Daily for up to 42 days postoperatively, at 6 months follow-up
  Painful areas are marked on a figure illustrating a human torso (both front and back are shown). The figure has predefined squares in order to standardize report.
Postoperative usage of analgesics | Daily for up to 42 days postoperatively, at 6 months follow-up
  Usage of analgesics is divided into non-opioid and opioid analgesics and into prescribed and as needed usage.
Postoperative usage epidural analgesia | Within 4 days postoperatively
  Usage of epidural analgesia is measured as both total and bolus infusion of epidural analgesics i millilitres (Ml)
Intensity of brush-evoked pain (mechanical allodynia) | At 6 weeks follow-up
  Any pain evoked by brush on the thorax (mechanical allodynia) is rated on 11-point numerical rating scale with the verbal anchors "No pain" and "Worst pain imaginable"
Intensity of brush-evoked discomfort (mechanical allodynia) | At 6 weeks follow-up
  Any discomfort evoked by brush on the thorax (mechanical allodynia) is rated on 11-point numerical rating scale with the verbal anchors "No discomfort" and "Worst discomfort imaginable"
Dysaesthesia | At 6 weeks follow-up
  Presence of dysaesthesia when stroking the skin on the thorax with a brush
Intensity of pinprick-evoked pain (mechanical dynamical hyperalgesia) | At 6 weeks follow-up
  Any pain evoked by pinprick (Von Frey) on the thorax (mechanical dynamical hyperalgesia) is rated on 11-point numerical rating scale with the verbal anchors "No pain" and "Worst pain imaginable"
Hypoalgesia (skin) | At 6 weeks follow-up
  Presence of hypoalgesia on the thorax is defined as a reduced response to pinprick (Von Frey)
Peri-incisional secondary hyperalgesia | At 6 weeks follow-up
  Negative difference between pressure pain thresholds (skinfold pinch) measured before surgery and at 6 weeks follow-up. Meassurements are made with a handheld pressure algometer 5 cm distal to the papilla
Generalized secondary hyperalgesia | At 6 weeks follow-up
  Negative difference between pressure pain thresholds (musculus quadriceps femoris) measured before surgery and at 6 weeks follow-up. Meassurements are made with a handheld pressure algometer in the quadriceps 10 cm above to the patella
Personality | At 6 months follow-up
  Response to Neuroticism, extraversion, openness, personality inventory - revised (NEO-PI-R) at 6 months follow-up compared to baseline
Pain Catastrophizing | At baseline, following coldpressor test, at 3 days postoperatively, at 6 months follow-up
  Responses to the Pain Catastrophizing Scale (PCS) compared to baseline
Anxiety | At baseline, following coldpressor test, at 3 days postoperatively, at 6 months follow-up
  Responses to the State-Trait Anxiety Inventory (STAI) compared to baseline
Depression | At baseline, at 3 days postoperatively, at 6 months follow-up
  Responses to the Beck's depression Inventory - second edition (BPI-II) compared to baseline
Emotions | At baseline, at 3 days postoperatively, at 6 months follow-up
  Responses to the Positive and Negative Affective Scale (PANAS) compared to baseline
Health-related Quality of life | At baseline, at 6 months follow-up
  Responses to the Short Form Health Survey (SF-36) compared to baseline
Self-esteem | At baseline, at 6 months follow-up
  Responses to the Rosenberg Self-esteem Scale (SES) compared to baseline
Qualitative dimension of pain | At baseline, following coldpressor test, at 3 days postoperatively, at 6 weeks follow-up, at 6 months follow-up
  Responses to the McGill Pain Questionnaire - short form (SF-MPQ) compared to baseline
Pain interference with daily life | At baseline, at 6 weeks follow-up, at 6 months follow-up
  Responses to the Brief Pain Inventory - short form (SF-BPI) compared to baseline
Course of pain | At 6 weeks follow-up, at 6 months follow-up
  Course of pain is defined as 1.) constant pain with few fluctuations, 2.) constant pain with breakthrough pain, 3.) Breakthrough pain without pain in between, 4.) Breakthrough pain with pain in between.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Vase, Cand.psyc, PhD, Study Chair — University of Aarhus; Mogens Pfeiffer-Jensen, MD, PhD, Study Chair — Department of Rheumatology, Aarhus University Hospital; Hans K Pilegaard, MD, Study Director — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby; Asbjørn M Drewes, Prof., MD, PhD, DMsc, Study Chair — Mech-Sense, Department of Gastroenterology, Aarhus University Hospital, Aalborg Hospital,; Vibeke E Hjortdal, Prof., MD, PhD, DMSc, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby; Kasper Grosen, PhD Student, Principal Investigator — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby
Locations (1):
- Department of Cardiothoracic and Vascular Surgery, Aarhus, Denmark